CLINICAL TRIAL: NCT06534567
Title: Association of Body Composition, Growth, and Maturation Status With Physical Activity and Adherence With Mediterranean Diet in Youth Triathletes
Brief Title: Body Composition, Growth, and Maturation of Triathletes
Status: Recruiting | Type: Observational
Sponsor: University of Alicante (Other)
Responsible Party: Principal Investigator, Jose Miguel Martinez Sanz, Associate Professor. Director of the Research Group on Applied Dietetics, Nutrition and Body Composition. Nursing Department. Faculty of Health Sciences. University of Alicante., University of Alicante
Other Study IDs: UA-2021-11-17
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Diet Habit; Body Weight Changes
MeSH Terms: conditions — Feeding Behavior; Body Weight Changes | interventions — Diet, Mediterranean; Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Male: Young male triathletes
  Interventions: Other: Mediterranean Diet; Other: Physical activity
- Female: Young female triathletes
  Interventions: Other: Mediterranean Diet; Other: Physical activity

INTERVENTIONS:
Other: Mediterranean Diet — Mediterranean diet adherence
Other: Physical activity — Physical activity level

SUMMARY:
The goal of this observational study is to determine if physical activity and the adherence to a Mediterranean diet have a relationship with body composition, growth, and maturation status in youth triathletes. The main question it aims to answer is:

• Is body composition (fat and muscle) determined primarily by growth and biological maturation or by physical activity and the Mediterranean diet in youth triathletes? Participants already have been evaluated in body composition, mediterranean diet adherence and practical of physical activity during 3 years.

DETAILED DESCRIPTION:
Triathlon is an individual, multidisciplinary and resistance sport with three stages: swimming, cycling and running, linked by two transitions. The importance of knowing body composition, eating patterns, level of physical activity and maturational state, will allow influence on training, increasing sports performance.

Regarding body composition and its relationship with performance, it has been observed that the greater the body fat, the lower the physical performance of triathletes. In each sport, athletes have different composition somatotypes. For triathlon, it is difficult to establish a specific somatotype, since it is a modality that encompasses three sports, among which the anthropometric characteristics of the athletes who practice them are not similar. In addition, since it is a relatively new category, there are not enough bibliographical references regarding anthropometry and body composition.

During biological maturation, there is an increase in the basal metabolic rate, so an optimal diet helps the growth process and improves the performance and recovery of athletes. Therefore, in the early stages of childhood and adolescence, adherence to the diet plays an important role in the acquisition of healthy lifestyles to determine an optimal state of health. The Mediterranean Diet model is associated with healthy eating habits, high levels of quality of life and physical benefits.

ELIGIBILITY:
Inclusion Criteria:

* Acceptation of informed consent by parents

Exclusion Criteria:

* No attendance to body composition evaluation
* Reporting less than 80% of assistance to physical activity sessions reported by trainer

Ages: 5 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: Young triathletes belonging to the ADESAVI triathlon club from the city of San Vicente del Raspeig (Spain)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Body Composition | 5 years
  Change in body composition (fat mass and muscle mass) by anthropometric evaluation

SECONDARY OUTCOMES:
Physical Activity Level | 5 years
  Low, moderate or high
Mediterranean Diet Adherence | 5 years
  Low, moderate or high
Biological Maturation Status | 5 years
  early, average or late maturers

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences. University of Alicante., San Vicent del Raspeig, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No
The data are available from the authors on request from the IP JMMS (josemiguel.ms@ua.es).

REFERENCES:
- [Background] Romero-Garcia D, Esparza-Ros F, Pico Garcia M, Martinez-Sanz JM, Vaquero-Cristobal R. Adherence to the Mediterranean diet, kinanthropometric characteristics and physical performance of young male handball players. PeerJ. 2022 Dec 1;10:e14329. doi: 10.7717/peerj.14329. eCollection 2022. PMID 36518299
- [Background] Albaladejo-Saura M, Vaquero-Cristobal R, Garcia-Roca JA, Esparza-Ros F. Influence of biological maturation status on selected anthropometric and physical fitness variables in adolescent male volleyball players. PeerJ. 2022 Apr 5;10:e13216. doi: 10.7717/peerj.13216. eCollection 2022. PMID 35402095
- [Background] Albaladejo-Saura M, Vaquero-Cristobal R, Gonzalez-Galvez N, Esparza-Ros F. Relationship between Biological Maturation, Physical Fitness, and Kinanthropometric Variables of Young Athletes: A Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2021 Jan 5;18(1):328. doi: 10.3390/ijerph18010328. PMID 33466291
- [Background] Mirwald RL, Baxter-Jones AD, Bailey DA, Beunen GP. An assessment of maturity from anthropometric measurements. Med Sci Sports Exerc. 2002 Apr;34(4):689-94. doi: 10.1097/00005768-200204000-00020. PMID 11932580
- [Background] Moran J, Sandercock G, Rumpf MC, Parry DA. Variation in Responses to Sprint Training in Male Youth Athletes: A Meta-analysis. Int J Sports Med. 2017 Jan;38(1):1-11. doi: 10.1055/s-0042-111439. Epub 2016 Oct 28. PMID 27793062